CLINICAL TRIAL: NCT02702713
Title: Investigation of the Effect of Daily Consumption of Bioactive Enriched Foods (BEF) on Biochemical and Anthropometric Markers of Metabolic Syndrome (MS)
Brief Title: Pivotal Assessment of the Effects of Bioactive on Health and Wellbeing. From Human Genome to Food Industry
Acronym: PATHWAY-27
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The funding agency set a mandatory deadline for the study in order to be able to conclude the project.
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Collaborators: Max Rubner-Institut (Unknown); University of Leeds (Other); Centre de Recherche en Nutrition Humaine d'Auvergne (Other Government); University of Bologna (Other)
Responsible Party: Principal Investigator, Luigi Ricciardiello, Associate Professor of Gastroenterology, University of Bologna, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 147/2015/U/Sper
Record Dates: First submitted 2016-02-18; First posted 2016-03-09 (Estimated); Last update posted 2017-12-02 (Actual); Status verified 2017-11

CONDITIONS: Metabolic Syndrome
Keywords: bioactive; enriched foods; anthocyanins (AC); beta-glucans (BG); docosahexaenoic acid (DHA)
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Dairy BEF + egg placebo + bakery placebo (Active Comparator): 200 subjects consuming every day for 12 weeks: 1 portion of Dairy BEF + 1 portion of Egg placebo + 1 portion of Bakery placebo
  Interventions: Dietary Supplement: Dairy BEF; Dietary Supplement: Bakery placebo; Dietary Supplement: Egg placebo
- Egg BEF + dairy placebo + bakery placebo (Active Comparator): 200 subjects consuming every day for 12 weeks: 1 portion of Egg BEF + 1 portion of Dairy placebo + 1 portion of Bakery placebo
  Interventions: Dietary Supplement: Egg BEF; Dietary Supplement: Bakery placebo; Dietary Supplement: Dairy placebo
- Bakery BEF + dairy placebo + egg placebo (Active Comparator): 200 subjects consuming every day for 12 weeks: 1 portion of Bakery BEF + 1 portion of Dairy placebo + 1 portion of Egg placebo
  Interventions: Dietary Supplement: Bakery BEF; Dietary Supplement: Dairy placebo; Dietary Supplement: Egg placebo
- All placebo (Placebo Comparator): 200 subjects consuming every day for 12 weeks: 1 portion of Egg placebo + 1 portion of Dairy placebo + 1 portion of Bakery placebo
  Interventions: Dietary Supplement: Bakery placebo; Dietary Supplement: Dairy placebo; Dietary Supplement: Egg placebo

INTERVENTIONS:
Dietary Supplement: Dairy BEF — Dairy BEF: Milkshake powder enriched with 250 mg of DHA and 3g beta-glucans
  Arms: Dairy BEF + egg placebo + bakery placebo
Dietary Supplement: Egg BEF — Egg BEF: Frozen pancakes enriched with 250 mg of DHA and 320 mg of anthocyanins
  Arms: Egg BEF + dairy placebo + bakery placebo
Dietary Supplement: Bakery BEF — Bakery BEF: Biscuits enriched with 250 mg of DHA and 320 mg of anthocyanins
  Arms: Bakery BEF + dairy placebo + egg placebo
Dietary Supplement: Bakery placebo — Bakery placebo: Biscuits without enrichment
  Arms: All placebo; Dairy BEF + egg placebo + bakery placebo; Egg BEF + dairy placebo + bakery placebo
Dietary Supplement: Dairy placebo — Dairy placebo: Milkshake powder without enrichment
  Arms: All placebo; Bakery BEF + dairy placebo + egg placebo; Egg BEF + dairy placebo + bakery placebo
Dietary Supplement: Egg placebo — Egg placebo: Frozen pancakes without enrichment
  Arms: All placebo; Bakery BEF + dairy placebo + egg placebo; Dairy BEF + egg placebo + bakery placebo

SUMMARY:
This is a multi-centre, randomised, double-blind, placebo-controlled, parallel-arm dietary intervention study. In total, 800 men and women at risk for Metabolic Syndrome (MS) will be recruited. Subjects will be eligible to the study if they present with two to four of the MS diagnostic criteria, at least one of them being:

* fasting triglycerides ≥150 mg/dL but ≤400 mg/dL OR
* HDL-cholesterol ≤50 mg/mL in women, ≤ 40mg/mL in men (with fasting triglycerides ≥110 mg/dL).

Each of the four recruiting centres will recruit 200 volunteers. Participants will be randomly assigned to one of four groups to receive either:

* Dairy BEF + egg placebo + bakery placebo
* Egg BEF + dairy placebo + bakery placebo
* Bakery BEF + dairy placebo + egg placebo
* Dairy, egg and bakery placebo

Participants will be required to consume all three of the allocated products each day for 12 weeks.

Eligible volunteers will be included and randomly allocated to one of the four groups. At baseline, 6 weeks and 12 weeks after inclusion, each participant will visit the recruiting centre for clinical and biochemical investigations. At 3 weeks and 9 weeks participants will complete questionnaires relating to their satisfaction with the food products, compliance to consumption of the study food products, and any gastrointestinal side effects or health-related adverse events that have occurred in the previous 3 weeks.

At each recruiting centre 40 participants will be required to take part in additional activities, these are: stool sample collection, adipose tissue aspiration, body composition analysis by dual energy x-ray absorptiometry (DEXA) and assessment of physical activity.

ELIGIBILITY:
Inclusion Criteria:

* subjects presenting with two to four diagnostic criteria for metabolic syndrome, at least one of them being elevated fasting triglycerides OR HDL-cholesterol ≤50 mg/mL in women, ≤ 40mg/mL in men (with fasting triglycerides ≥110 mg/dL).

Exclusion Criteria:

* subjects with five clinical criteria for metabolic syndrome
* Regular drug therapy with impact on serum lipids;
* Diabetes (fasting glucose > 1.26 g/L, or anti-diabetic treatment);
* Celiac disease, lactose intolerance, allergy to milk or egg proteins;
* Antibiotic treatment within the last 3 months;
* Recent history of cancer or cancer treatment (less than 2 years);
* Active or recently diagnosed intestinal malabsorption;
* Diagnosis of organ failure
* Familial dyslipidemia (TG ≥ 4.5 mmol/l or 400 mg/dl);
* Illegal drug use or chronic alcoholism or smoking;
* Intensive physical exercise (≥ 5 hour/week);
* Consumption of nutritional supplements containing DHA, BG or AC;
* History of allergy or intolerance to any components used in BEF;
* Women who are pregnant or lactating;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 325 (Actual)
Dates: Start 2016-02; Primary Completion 2017-10-20 (Actual); Study Completion 2017-10-20 (Actual)

PRIMARY OUTCOMES:
Triglycerides blood levels (mg/dl) | Baseline and 12 weeks
  Change from baseline in triglycerides blood levels after 12 weeks of consumption of foods enriched with DHA, alone or in combination with AC or BG, in subjects at risk for or affected by MS.
HDL-cholesterol blood levels (mg/dl) | Baseline and 12 weeks
  Change from baseline in HDL-cholesterol blood levels after 12 weeks of consumption of foods

SECONDARY OUTCOMES:
Blood glucose (mg/dl). | Baseline and 12 weeks
  Change from baseline in blood glucose levels after 12 weeks of consumption of foods enriched with DHA, alone or in combination with AC or BG, in subjects at risk for or affected by MS.
Blood pressure (mmHg) | Baseline and 12 weeks
  Change from baseline in blood pressure after 12 weeks of consumption of foods enriched with DHA, alone or in combination with AC or BG, in subjects at risk for or affected by MS.
Waist circumference (cm). | Baseline and 12 weeks
  Change from baseline in waist circumference after 12 weeks of consumption of foods enriched with DHA, alone or in combination with AC or BG, in subjects at risk for or affected by MS.
Urinary food metabolite levels (parts per millions). | Baseline and 12 weeks
  Changes from baseline in urinary food metabolite levels, after 12 weeks of consumption of foods enriched with DHA, alone or in combination with AC or BG, in subjects at risk for or affected by MS.
Fecal microbiota composition (analysis of principal coordinates - PCOA) | Baseline and 12 weeks
  Changes in fecal bacterial composition and diversity will be determined at baseline and after 12 weeks of consumption of foods enriched with DHA, alone or in combination with AC or BG, in subjects at risk for or affected by MS. The predominant microbial community and specific functional groups will be characterized by next-generation sequencing (NGS) of the 16S rDNA gene. The interindividual differences in the composition of the intestinal microbiota (beta-diversity) will be evaluated with the analysis of principal coordinates (PCOA). Appropriate statistical analysis will be performed to evaluate significant differences in the relative abundance of the microbial groups of intestinal microbiota between different groups of subjects.
Fecal Short Chain Fatty Acids (parts per million). | Baseline and 12 weeks
  Change from baseline in production/uptake in the stool of Short Chain Fatty Acids, after 12 weeks of consumption of foods enriched with DHA, alone or in combination with AC or BG, in subjects at risk for or affected by MS.
Dna methylation levels (%). | Baseline and 12 weeks
  To test whether lymphocytes may be useful as a surrogate for adipose tissue to detect changes in DNA methylation and gene expression, genome-wide methylation differences will be performed in parallel in lymphocytes and fat cells from baseline and after 12 weeks of consumption of foods enriched with DHA, alone or in combination with AC or BG, in subjects at risk for or affected by MS. Expression of affected genes will be evaluated by qRT-PCR.
Serum Hemoglobin A1c (HbA1c) levels (%) | Baseline and 12 weeks
  Change from baseline in HbA1c levels, after 12 weeks of consumption of foods enriched with DHA, alone or in combination with AC or BG, in subjects at risk for or affected by MS.
Homeostasis Model Assessment (HOMA) Index levels. | Baseline and 12 weeks
  Change from baseline in Homeostasis Model Assessment Index levels, after 12 weeks of consumption of foods enriched with DHA, alone or in combination with AC or BG, in subjects at risk for or affected by MS.
Fecal metabolite levels (parts per millions). | Baseline and 12 weeks
  Change from baseline in food metabolite levels in the stools after 12 weeks of consumption of foods enriched with DHA, alone or in combination with AC or BG, in subjects at risk for or affected by MS.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Bordoni, MD, Study Director — Department of Agro-Food Sciences and Technologies, University of Bologna
Locations (4):
- Centre de Récherche en Nutrition Humaine d'Auvergne, Clermont-Ferrand, Auvergne, France
- Max Rubner-Institut, Karlsruhe, Baden-Wurttemberg, Germany
- University of Bologna, Department of Medical and Surgical Sciences and Azienda Ospedaliero Universitaria di Bologna, Policlinico S.Orsola-Malpighi, Bologna, BO, Italy
- University of Leeds, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Individual case report forms are available to collect study data into electronic form from all the recruiting centres. A central electronic database has been elaborated to capture, validate and manage the entered data by means of a variety of edit checks (e.g., subjecting the data to range checks, valid value checks, cross-checks, and manual review) that provide feedback to those entering/providing the data.

REFERENCES:
- See also: Pathway-27 website — http://www.pathway27.eu/